CLINICAL TRIAL: NCT02376088
Title: Characteristics of Islet β-cell Functions in Chinese Patients With Graves' Disease
Status: Completed | Type: Observational
Sponsor: Weikai Hou (Other)
Responsible Party: Sponsor-Investigator, Weikai Hou, Professor, Qilu Hospital of Shandong University
Organization: Qilu Hospital of Shandong University (Other)
Other Study IDs: GD-003
Record Dates: First submitted 2015-02-18; First posted 2015-03-03 (Estimated); Last update posted 2015-03-03 (Estimated); Status verified 2015-02

CONDITIONS: Graves Disease
MeSH Terms: conditions — Graves Disease | interventions — Methimazole

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (7):
- GA1: subjects from coastal areas who initiated Methimazole treatment for the first time on enrollment
  Interventions: Drug: Methimazole
- GA2: subjects from coastal areas who were under Methimazole treatment and with an elevated TH level
  Interventions: Drug: Methimazole
- GA3: subjects from coastal areas who were under Methimazole treatment and with a normal TH level
  Interventions: Drug: Methimazole
- GB1: subjects from non-coastal areas who initiated Methimazole treatment for the first time on enrollment
  Interventions: Drug: Methimazole
- GB2: subjects from non-coastal areas who were under Methimazole treatment and with an elevated TH level
  Interventions: Drug: Methimazole
- GB3: subjects from non-coastal areas who were under Methimazole treatment and with a normal TH level
  Interventions: Drug: Methimazole
- NC: age-matched healthy checkup subjects

INTERVENTIONS:
Drug: Methimazole — All enrolled subjects with GD were treated with methimazole. The initial dose for the GA1 and GB1 sungroups were 30 mg/d (10 mg, tid), TH levels were tested every month, and the dose was titrated accordingly over a period of 2-3 months, the dose was then decreased to 15-20 mg/d and thyroid function was monitored periodically until it eventually reached the maintenance dose of 2.5 mg-5.0 mg/d. The dose and adjustment method for GA2 and GB2 were the same with GA1 and GB1, while the dose for GA3 and GB3 was gradually decreased to 2.5-5.0 mg/d. All subjects underwent a treatment course over a period of 6 months.
  Other Names: Thyrozol
  Groups: GA1; GA2; GA3; GB1; GB2; GB3

SUMMARY:
Patients with GD often present with glucose dysregulation, which, according to most studies, is associated with islet β-cell dysfunctions, enhanced gluconeogenesis and insulin resistance (IR). Current studies focus mainly on IR, and a few that investigate islet β-cell functions show inconsistent results. This study examined the characteristics of glucose dysregulation in Chinese patients with GD, and furthermore evaluated the effects of thyroid dysfunction on islet β-cell functions and subsequently the carbohydrate metabolism.

DETAILED DESCRIPTION:
Thyroid dysfunction is closely associated with glucoregulation. Carbohydrate metabolism can be affected with decreased levels of thyroid hormone (TH), even more so with an elevated TH level. Epidemiological data shows that 2%-57% of patients with Graves' Disease (GD) present with glucose dysregulation, which might also be related to the changes in islet β-cell functions in patients with GD. The incidence of GD has comparable variations geographically, with possibly different underlying mechanisms, such as an excessive intake of iodine resulting in an aggravation of autoimmune reactions from thyroid and consequently an increment in incidence of GD. The same might also be true in glucoregulation and islet β-cell functions in patients with GD. This study aims to examine the characteristics of glucoregulation and islet β-cell functions in patients with GD in different areas of China, using early-phase insulin secretion index (△I30/△G30), glucose area under curve(GAUC) and insulin area under curve(INSAUC).

ELIGIBILITY:
Inclusion Criteria:

* Patients with Graves Disease
* Age-matched healthy checkup subjects

Exclusion Criteria:

* Patients with a medical history of diabetes, pancreatitis and other related conditions and positive family histories as well as medication history of glucocorticoid and anti-diabetic agents

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: A total of 283 outpatients, aged 22 to 55 years old(mean age 39±4 years), of whom 41 were male and 242 were female (M/F=1/5.90), were enrolled for the study from Qilu Hospital of Shandong University and Shandong Jiaotong Hospital between June, 2011 and June, 2014. An additional 45 age-matched healthy checkup subjects were included in the normal control group (NC). Patients with a medical history of diabetes, pancreatitis and other related conditions and positive family histories as well as medication history of glucocorticoid and anti-diabetic agents were excluded.
Sampling Method: Non-Probability Sample
Enrollment: 328 (Actual)
Dates: Start 2011-06; Primary Completion 2014-06 (Actual); Study Completion 2014-06 (Actual)

PRIMARY OUTCOMES:
change from baseline blood glucose at 6 months | at the day of the subject's enrollment into the study(baseline) and at 6 months after the enrollment
change from baseline insulin at 6 months | at the day of the subject's enrollment into the study(baseline) and at 6 months after the enrollment
change from baseline thyroid hormone at 6 months | at the day of the subject's enrollment into the study(baseline) and at 6 months after the enrollment
change from baseline urine iodine concentration at 6 months | at the day of the subject's enrollment into the study(baseline) and at 6 months after the enrollment